CLINICAL TRIAL: NCT02795897
Title: Genomic Translation for Amyotrophic Lateral Sclerosis Care
Acronym: GTAC
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: ALS Association (Other); Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: AAAQ7026
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: ALS
Keywords: genetics; genomics; amyotrophic lateral sclerosis (ALS); primary lateral sclerosis (PLS); progressive muscular atrophy (PMA); motor neuron disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA and Peripheral blood mononuclear cells (PBMCs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to look for abnormal genes and gene expression profiles that help determine why a person develops amyotrophic lateral sclerosis (ALS) and related motor neuron diseases (MND) and why their symptoms present and progress with a particular pattern.

DETAILED DESCRIPTION:
In all patients, ALS/MND is caused by the progressive death of motor neurons. However, every patient is affected differently. Some develop symptoms in their 80's while others get sick in adolescence. Swallowing/speech are affected first in some patients, but most have weakness in their hands or feet at onset. Some individuals show very rapid progression, even as others live for decades. Finally, some patients have loss of mainly motor neurons in the brain (as in primary lateral sclerosis), while others lose mainly lower motor neurons in the spinal cord and brain stem (as in progressive muscular atrophy). Research has uncovered a few genetic factors that contribute to the variability of ALS/MND. For example, mutations in the superoxide dismutase 1 (SOD1) gene makes onset in the legs more likely and decreases the chance of developing dementia. Conversely, having a mutated C9ORF72 gene makes dementia much more likely. Uncovering additional factors causing ALS variability is an important research priority and is likely to provide clues about how to better diagnose and treat the disease.

This study is called "Genomic Translation for ALS Care" (GTAC). The investigators will analyze the genome and gene expression patterns of people with ALS/MND and carry out research on that data, finding insights that the investigators hope will translate into better care for ALS/MND patients.

ELIGIBILITY:
Inclusion Criteria:

Study participants meeting all of the following criteria will be eligible for enrollment in GTAC:

1. Men or women of any race or ethnicity aged 18 or older
2. Diagnosis of familial or sporadic ALS (definite, probable, or possible according to El Escorial Criteria, Appendix 1), or those with primary lateral sclerosis or progressive bulbar/muscular atrophy forms of motor neuron disease. All-comers with ALS/MND should be enrolled without regard to familial vs sporadic or gene mutation status (i.e. participants with known gene mutations should still be enrolled), or phenotype.
3. Capable of providing informed consent and following study procedures (in the case that a subject lacks the ability to provide informed consent, informed consent will be sought from the subject's surrogate representative).
4. Willing to return to clinic site (or another participating center) for follow-up care.

Exclusion Criteria:

Study participants meeting any of the following criteria during screening evaluation will be excluded from enrolling in GTAC:

1. Invasive ventilation (i.e. tracheostomy) in place.
2. Non-invasive ventilation dependent (defined as >22 hours per day)
3. Pregnancy.
4. Known Human Immunodeficiency Virus (HIV) , chronic Hepatitis B, or Hepatitis C (because cells will be frozen down for future cell line generation).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ALS (meeting El Escorial criteria for definite, probable or possible ALS), or primary lateral sclerosis or progressive bulbar/muscular atrophy.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Correlation of DNA genotype with ALS phenotypes | 36 months
  Because subjects are followed over their entire disease course and undergo whole genome sequencing of their DNA, this project will study the distinct features (progression and particular symptoms) of subjects with and without mutations in already known ALS genes.
Correlation of gene expression in blood with ALS phenotypes | 36 months
  Because subjects are followed over their entire disease course and undergo gene expression profiling on their blood sample, this project will study the distinct features (progression and particular symptoms) of subjects with different types of gene expression profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Harms, MD, Principal Investigator — Columbia University
Locations (14):
- United States (13):
  - Cedar Sinai Medical Center, Los Angeles, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Univeristy of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Oregon Health & Sciences University, Portland, Oregon
  - Penn State College of Medicine, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Houston Methodist Neurological Institute, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- The University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The investigators intend to share DNA, sequencing data, and phenotypic data broadly. Participants will be consented for sharing of GTAC data and samples with the Northeast ALS Consortium (NEALS) repository, with others carrying out ALS/MND research (including other consortia), for biomedical research in general (including use as controls and use by for-profit companies), and with Biogen Idec. Additionally, GTAC has plans to share coded genomic and clinical data with Database of Genotypes and Phenotypes (dbGaP) and a ALS/MND consortium for genomic discovery (ASLGEN). This includes sharing of genetic and phenotypic data with Biogen Idec, a pharmaceutical company that is partnering with GTAC to fund the sequencing of samples.
Time Frame: At the end of the study.
Access Criteria: The investigators intend to share DNA, sequencing data, and phenotypic data with the NEALS repository and Biogen Idec. Coded genomic and clinical data will be shared with dbGaP and ASLGEN.